CLINICAL TRIAL: NCT06552637
Title: RECOVER-HF - RandomizEd, Multi-Center, Double-Blinded Study of SynchrOnized Diaphragmatic Stimulation (SDS) for ImproVEment of Symptomatic Reduced Ejection Fraction Heart Failure
Brief Title: Synchronized Diaphragmatic Stimulation in Symptomatic Heart Failure
Acronym: RECOVER-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VisCardia Inc. (Industry)
Collaborators: Clinical Accelerator (Industry); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VisCardia H03_22
Record Dates: First submitted 2024-08-06; First posted 2024-08-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure; Heart Disease; Synchronized Diaphragmatic Stimulation; Implantable Heart Failure Device Therapy
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Initial randomization into Control and Therapy arms for 6 month primary endpoints, afterwards crossover of Control arm into Therapy arm for 12 month secondary endpoints.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator and care provider blinded to device programming, therapy imperceptible to patient, data analysis through independent entities
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device and Medical Management (Experimental): * Subjects will be implanted with the VisONE System programmed to deliver SDS (Therapy On) and receive optimal, stable, Guideline Directed Medical Therapy (GDMT) for heart failure (American Heart Association [AHA] / American College of Cardiology [ACC] guidelines) including those drugs to be determined by the subject's physician
  * Assigned Interventions:
    * Device: VisONE System (SDS)
    * Drug: Medical Management
  Interventions: Device: Synchronized Diaphragmatic Stimulation
- Medical Management (Sham Comparator): * Subjects will be implanted with the VisONE System programmed not to deliver SDS (Therapy Off) and receive optimal, stable, Guideline Directed Medical Therapy (GDMT) for heart failure (American Heart Association [AHA] / American College of Cardiology [ACC] guidelines) including those drugs to be determined by the subject's physician
  * Assigned Interventions:
    * Drug: Medical Management
  Interventions: Device: Synchronized Diaphragmatic Stimulation

INTERVENTIONS:
Device: Synchronized Diaphragmatic Stimulation — Implantable Pulse Generator system providing cardiac-gaited stimulation of the diaphragm and thereby influence cardiovascular properties relevant in heart failure.
  Other Names: Asymptomatic Diaphragmatic Stimulation; SDS; ADS; VisONE SDS

SUMMARY:
RECOVER HF is a clinical study designed to evaluate the safety and efficacy of Synchronized Diaphragmatic Stimulation delivered using the VisONE System in the treatment of patients with heart failure.

DETAILED DESCRIPTION:
Symptomatic Diaphragmatic Stimulation (SDS) is a novel extra-cardiac device for patients who have symptomatic heart failure. Elevated intracardiac pressures are the hallmark of heart failure (HF) and a key pathological driver of disease progression and limited exertional capacity. The degree of cardiac pressure elevation is determined by preload, afterload, and pericardial restraint. The pericardium restrains the heart, and the degree of restraint is determined by the pericardial structure itself and the intrathoracic pressure. This aspect of HF pathophysiology is among the fundamental drivers behind the SDS therapy concept. SDS induces a temporal modulation of intrathoracic pressure.. When synchronized with the cardiac cycle, SDS may improve cardiac filling, cardiovascular pressure conditions, and cardiac performance

RECOVER HF is a prospective, randomized, doubled-blinded study of Synchronized Diaphragmatic Stimulation (SDS) delivered in an imperceptible manner in subjects with heart failure defined as New York Heart Association (NYHA) functional class II/III, left-ventricular ejection fraction (LVEF) <=40%, and QRS duration <=130ms despite receiving the appropriate heart failure guideline directed medical therapy (GDMT). All subjects will receive an implanted VisONE System. Two-weeks post implant subjects will be randomized in a 1:1 ratio into a SDS therapy active or control (SDS therapy inactive) arm with both arms receiving GDMT. At 6 months the control arm will have SDS therapy activated with all patients receiving therapy and GDMT throughout the remainder of the study period. The study will be conducted at up to 30 investigational sites in the United States and several outside the U.S. These centers will enroll subjects with the goal of randomizing approximately 270 subjects who meet the entry criteria.

ELIGIBILITY:
Inclusion Criteria:

* NYHA classes II/III on optimal Guideline Directed Medical Therapy (GDMT)
* QRS duration ≤ 130 ms
* EF≤ 40%

Exclusion Criteria:

* Baseline 6 minute walk test > 500 meters or < 200 meters
* NT-proBNP< 250 if on loop diuretics, or NT-proBNP < 500 if not on loop diuretics
* Supine resting heart rate > 140 bpm
* Systolic blood pressure < 80 mmHg or > 170 mmHg
* Serum creatinine > 2.5 mg/dL
* Serum hepatic function 3x ULN
* Any of the following within the previous 3 months: unstable angina, AMI, CABG, PTCA, CVA/TIA, persistent AF (> 24 hours), symptomatic NSVT or DCCV
* Any inotropic drug treatment within the previous 3 months
* Bradycardia (heart rate < 50 beats/min), atrial arrhythmias with rates > 100 beats/min, sustained ventricular tachycardia or frequent ventricular ectopy >10% present during screening
* Significant uncontrolled symptomatic bradyarrhythmia, atrial fibrillation, unstable ventricular arrhythmias or frequent ventricular ectopy > 10% documented within the previous 3 months
* Reversible non-ischemic cardiomyopathy
* Valvular disease requiring intervention within the next 12 months or presence of significant valve disease as determined by the site cardiologist as:

  1. Greater than mild mitral valve stenosis
  2. Greater than moderate mitral valve regurgitation
  3. Greater than mild tricuspid valve stenosis
  4. Greater than moderate-severe tricuspid valve regurgitation
  5. Greater than moderate aortic stenosis
  6. Greater than moderate aortic regurgitation
  7. Greater than mild-moderate pulmonic stenosis
  8. Greater than moderate pulmonic regurgitation
* Severe primary pulmonary disease, including pulmonary arterial hypertension. PAP sys >70 mmHg at rest
* Severe COPD, other respiratory or lung diseases where FEV < 50%
* Presence of more than small pleural effusion or history of pleural drainage within the previous 6 months
* Known history of diaphragmatic paralysis or suspicion confirmed by unilateral or bilateral elevation of the diaphragm on chest x-ray
* Pericardial disease
* Diabetic neuropathy
* Existing diaphragmatic stimulation for respiration assist
* Present LVAD, Baroreflex Activation Therapy, Cardiac Contractility Modulation or interatrial shunt devices; temporary mechanical cardiac assist devices (current or within the previous 3 months); or CRT that is indicated or implanted and functional
* Contraindications to laparoscopic access to the diaphragm, as determined by the implanting physician
* Known intra-abdominal pathology which could increase the risk of laparoscopic access to the diaphragm.
* Previous open laparotomy within 1 year
* Previous thoracic or abdominal organ transplant
* Drug induced immuno-suppression
* Body mass index > 40
* Enrollment in a concurrent investigation / clinical study
* Having a life expectancy of <1 year due to any condition
* Pregnant or planning a pregnancy during the study period
* Known allergies to implantable device materials
* History of systemic infection requiring the use of intravenous antibiotics within the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricular End-Systolic Volume (LVESV) | 6 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger percent improvement in LVESV at 6 months post-randomization from baseline than medical management alone.
Six Minute Hall Walk (6MHW) | 6 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger improvement in 6MHW at 6 months post-randomization from baseline than medical management alone.
Minnesota Living with Heart Failure quality of Life Score (MLWHF QOL) | 6 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger improvement in MLWHF QOL at 6 months post-randomization from baseline than medical management alone.
Major Adverse Respiratory and Cardiovascular Events (MARCE) | 6 months
  To demonstrate the safety of the VisONE System by analyzing Major Adverse Respiratory and Cardiovascular Events (MARCE) occurring within 6 months post implant for the rate, severity and association with the device or procedure (goal >70% freedom):
  * Cardiovascular Death
  * Stroke
  * Cardiac Arrest
  * Interaction with cardiac rhythm device requiring permanent termination of SDS therapy
  * Acute Heart Failure Decompensation
  * Infection requiring device/lead explant
  * Diaphragmatic dysfunction leading to a clinically significant reduction is respiratory function
  * Inadequate SDS therapy delivery requiring surgical intervention
  * Injury to abdominal organs requiring surgical intervention
  * Pneumothorax
  * Hemothorax

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) | 6 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger improvement in LVEF at 6 months post-randomization from baseline than medical management alone.
N-Terminal Pro Brain Natriuretic Peptide (NT-proBNP) | 6 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger reduction in NT-proBNP (log-10 transformed) at 6 months post-randomization from baseline than medical management alone.
Left ventricular End-Systolic Volume (LVESV) | 12 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger percent improvement in LVESV at 12 months post-randomization from baseline than medical management alone.
Six Minute Hall Walk (6MHW) | 12 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger improvement in 6MHW at 12 months post-randomization from baseline than medical management alone.
Minnesota Living with Heart Failure quality of Life Score (MLWHF QOL) | 12 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger improvement in MLWHF QOL at 12 months post-randomization from baseline than medical management alone.
Left Ventricular Ejection Fraction (LVEF) | 12 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger improvement in LVEF at 12 months post-randomization from baseline than medical management alone.
N-Terminal Pro Brain Natriuretic Peptide (NT-proBNP) | 12 months
  To demonstrate that treatment with the VisONE System (SDS) plus GDMT results in a larger reduction in NT-proBNP (log-10 transformed) at 12 months post-randomization from baseline than medical management alone.

CONTACTS AND LOCATIONS:
Overall Officials: Lee R Goldberg, MD, Principal Investigator — University of Pennsylvania